CLINICAL TRIAL: NCT03256877
Title: Detecting Transitional Cell Carcinoma From Haematuria: A Study of Urinary Tissue Factor
Brief Title: Detecting Transitional Cell Carcinoma From Haematuria
Acronym: TransTuFo
Status: Completed | Type: Observational
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: C-Term Diagnostics Ltd (Unknown); Hull York Medical School (Unknown)
Responsible Party: Sponsor
Other Study IDs: R2006
Record Dates: First submitted 2017-08-15; First posted 2017-08-22 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Transitional Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: Patients with haematuria.

SUMMARY:
To validate ELISAs for the detection of urinary tissue factor (TF) in patients suspected of having bladder cancer.

DETAILED DESCRIPTION:
The effective diagnosis of transitional cell carcinoma (TCC), the most common form of bladder cancer, is often quite challenging, due to a lack of disease-specific symptoms. Detecting TCC early is crucial to increase the chances of a cure. Cystoscopy, which is currently the standard test used for urothelial cancer diagnosis, is an invasive and relatively expensive procedure but, while several potential markers in urine have been studied with the goal of replacing cystoscopy, no urinary marker alone or in combination with others has shown sufficient accuracy.

In this study, levels of tissue factor (TF) isoforms will be measured by ELISA in urine samples collected from patients referred to the haematuria clinic with visible or microscopic haematuria. These values will be linked to the subsequent diagnosis of each patient, and used to assess the accuracy of the ELISAs in detecting TCC when compared to standard cystoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving written informed consent
* Age ≥18 years
* Referral to haematuria clinic (gross or microscopic haematuria)

Exclusion Criteria:

* Inability to provide written informed consent
* Previous radiotherapy to the bladder (e.g. prostate cancer)
* Active urinary tract infection (Patients may be re-approached at later opportunity when urinary infection is cleared and haematuria persists)
* Current or planned treatment with neoadjuvant chemotherapy or radiotherapy
* Other known malignant condition, either active or in complete remission ≤5 years
* HIV, hepatitis C, or any other known communicable disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited from all patients referred to the haematuria clinic due to gross (visible) haematuria or findings on routine urinalysis suggestive of microscopic haematuria. These patients will be undergoing routine investigative cystoscopy on suspicion of urothelial cancer.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2018-05-28 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
Specificity and sensitivity of the ELISAs when compared to standard cystoscopy. | Outcome measure will be assessed by 6 months after trial completion.
  To examine the specificity and sensitivity of the ELISAs, compared to cystoscopy, in urine samples from patients presenting with gross or microscopic haematuria. The assays will provide measurements of the TF isoform concentrations present in patient urine samples, and the information on a subsequent diagnosis (or non-diagnosis) of a urothelial cancer will be obtained through reference to medical records.

SECONDARY OUTCOMES:
Positive and negative predictive values of the ELISAs when compared to standard cystoscopy. | Outcome measure will be assessed by 6 months after trial completion.
  To determine the positive and negative predictive values of the ELISAs, compared to cystoscopy, in urine samples from patients presenting with gross or microscopic haematuria.

CONTACTS AND LOCATIONS:
Locations (1):
- Castle Hill Hospital, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: No